CLINICAL TRIAL: NCT02751970
Title: Randomized Clinical Trial of the Effect of Different Categories of Adhesive System
Brief Title: Clinical Trial of the Effect of Different Categories of Adhesive System
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad de Valparaiso (Other)
Collaborators: Universidade Estadual de Ponta Grossa (Other)
Responsible Party: Principal Investigator, Issis luque, Professor, Universidad de Valparaiso
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CB027-2014
Record Dates: First submitted 2016-04-21; First posted 2016-04-26 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Dental Caries
Keywords: Dental adhesive; adhesive systems; Dental Restoration Failure
MeSH Terms: conditions — Dental Caries | interventions — SE 1-step Futurabond M

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 3 step ER & Dental restoration (Active Comparator): Dental restoration with etching the dental substrates 35% phosphoric acid, followed by the application of a primer and subsequently an adhesive resin.
  Interventions: Procedure: Dental restoration; Procedure: 3 step ER
- 2 step ER & Dental restoration (Experimental): Dental restoration with etching the dental substrates 35% phosphoric acid, followed by the application of an adhesive/primer step.
  Interventions: Procedure: Dental restoration; Procedure: 2 step ER
- 2 step SE & Dental restoration (Active Comparator): Dental restoration with etching the dental substrates with acidic primer, followed by the application of adhesive resin.
  Interventions: Procedure: Dental restoration; Procedure: 2 step SE
- 1 step SE & Dental restoration (Experimental): Dental restoration with etching and infiltrate the dental substrates with acidic primer/adhesive system.
  Interventions: Procedure: Dental restoration; Procedure: 1 step SE

INTERVENTIONS:
Procedure: Dental restoration — Methacrylate resins will be used to complement the cavity restoration after of adhesive procedure
  Other Names: Dental resin restoration
Procedure: 3 step ER — Enamel and dentin will be conditioning with 35% phosphoric acid, then applied primer, and then applied adhesive resin.
  Arms: 3 step ER & Dental restoration
Procedure: 2 step ER — Enamel and dentin will be conditioning with 35% of phosphoric acid, then applied primer/adhesive resin.
  Arms: 2 step ER & Dental restoration
Procedure: 2 step SE — Enamel and dentin will be conditioning with acidic primer, then applied primer/adhesive resin.
  Arms: 2 step SE & Dental restoration
Procedure: 1 step SE — Enamel and dentin will be conditioning with acidic primer/adhesive resin.
  Arms: 1 step SE & Dental restoration

SUMMARY:
This study aims to evaluate the clinical effectiveness of contemporary resin-based adhesive systems by retention rate of resin restorations placed in non carious cervical lesions with four different adhesive strategies: 3 and 2 steps etch-and-rinse adhesive system, 2 and 1 step self-etch adhesive systems.

DETAILED DESCRIPTION:
The etch-and-rinse (3 and 2 steps) and self-etch (1 and 2 steps) adhesive systems allow the bond between the resins restorations with the dental substrates, but they have mechanism of action different.

The success of resin composite restorations is reliant upon adhesion to the underlying tooth via adhesive systems. The mechanism of adhesion to enamel and dentine could be involved for one hand, the etching the substrates with 30-40% phosphoric acid, followed by the application of a primer and subsequently an adhesive resin 3 steps etch-and- rinse approach or 2 steps when to combine the primer and adhesive into one bottle. For another hand, the self- etch systems with acid monomers in their primer, allow conditioning the surface without phosphoric acid step. So, they consist of either a self-etching primer accompanied by an adhesive resin applied as a subsequent step (2 steps) or a self-etch adhesive, which does not require a separate primer (1 step).

ELIGIBILITY:
Inclusion Criteria:

* Good general health,
* Patients with acceptable oral hygiene level,
* Patients with at least 20 teeth under occlusion.
* Patients with at least four non-carious cervical lesions in four different teeth
* Patients with maximum of eight lesions that needed to be restored.
* These lesions had to be non-carious, non-retentive, deeper than 1 mm, and involve both the enamel and dentin of vital teeth without mobility.

Exclusion Criteria:

* Patients with extremely poor oral hygiene,
* Patients with severe or chronic periodontitis,
* Patients with heavy bruxism habits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 185 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-05 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Secondary caries | one year
  Secondary caries near and/or associated of the dental restorations
Retention rate | one year
  retention rate of the dental restorations

SECONDARY OUTCOMES:
Marginal integrity | one year
  marginal integrity of the dental restorations
Marginal discoloration | one year
  Marginal discoloration of the dental restorations
post-operative sensitivity | one year
  dentin post-operative sensitivity

CONTACTS AND LOCATIONS:
Overall Officials: Issis Luque, professor, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Universidad Valparaiso, Valparaíso, Región de Valparaíso, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chee B, Rickman LJ, Satterthwaite JD. Adhesives for the restoration of non-carious cervical lesions: a systematic review. J Dent. 2012 Jun;40(6):443-52. doi: 10.1016/j.jdent.2012.02.007. Epub 2012 Feb 18. PMID 22353603
- [Background] Eliguzeloglu Dalkilic E, Omurlu H. Two-year clinical evaluation of three adhesive systems in non-carious cervical lesions. J Appl Oral Sci. 2012 Mar-Apr;20(2):192-9. doi: 10.1590/s1678-77572012000200012. PMID 22666836
- [Background] Kurokawa H, Miyazaki M, Takamizawa T, Rikuta A, Tsubota K, Uekusa S. One-year clinical evaluation of five single-step self-etch adhesive systems in non-carious cervical lesions. Dent Mater J. 2007 Jan;26(1):14-20. doi: 10.4012/dmj.26.14. PMID 17410888
- [Background] Scotti N, Comba A, Gambino A, Manzon E, Breschi L, Paolino D, Pasqualini D, Berutti E. Influence of operator experience on non-carious cervical lesion restorations: Clinical evaluation with different adhesive systems. Am J Dent. 2016 Feb;29(1):33-8. PMID 27093774
- [Background] Moosavi H, Kimyai S, Forghani M, Khodadadi R. The clinical effectiveness of various adhesive systems: an 18-month evaluation. Oper Dent. 2013 Mar-Apr;38(2):134-41. doi: 10.2341/12-110-CR. Epub 2012 Aug 23. PMID 22917442
- [Background] Heintze SD, Blunck U, Gohring TN, Rousson V. Marginal adaptation in vitro and clinical outcome of Class V restorations. Dent Mater. 2009 May;25(5):605-20. doi: 10.1016/j.dental.2008.11.004. Epub 2009 Jan 14. PMID 19147216
- [Background] Peumans M, Kanumilli P, De Munck J, Van Landuyt K, Lambrechts P, Van Meerbeek B. Clinical effectiveness of contemporary adhesives: a systematic review of current clinical trials. Dent Mater. 2005 Sep;21(9):864-81. doi: 10.1016/j.dental.2005.02.003. PMID 16009415
- [Background] Van Landuyt KL, Mine A, De Munck J, Jaecques S, Peumans M, Lambrechts P, Van Meerbeek B. Are one-step adhesives easier to use and better performing? Multifactorial assessment of contemporary one-step self-etching adhesives. J Adhes Dent. 2009 Jun;11(3):175-90. PMID 19603581
- [Background] van Dijken JW. Clinical evaluation of three adhesive systems in class V non-carious lesions. Dent Mater. 2000 Jul;16(4):285-91. doi: 10.1016/s0109-5641(00)00019-1. PMID 10831784